CLINICAL TRIAL: NCT05966558
Title: Cesarean Section Scar Niche: The Impact on Assisted Reproductive Technology Outcome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Rana Nabil Mohamed Attia, Assistant lecturer of obstetrics and gynaecology, Zagazig University
Other Study IDs: 9385-22-3-2022
Record Dates: First submitted 2021-01-20; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Cesarean Section Niche Impact on ART
Keywords: Cesarean Section niche

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
the presence of cesarean section niche has adverse effects on success of ART outcome

DETAILED DESCRIPTION:
A common finding by ultrasound in secondary infertility patients with previous cesarean sections is the presence of niche, which is formally defined as an indentation of the uterine myometrium of at least 2 mm at the site of the caesarean scar. The most common symptom of niche is abnormal uterine bleeding, other symptoms include dysmenorrhea, chronic pelvic pain, dyspareunia, and sub-fertility/infertility.

It has been reported that a niche can reduce the chances of embryo implantation and may lead to spontaneous miscarriages if the implantation is close to or in the niche. The presence of a niche may render the actual embryo transfer procedure technically more difficult, and clinicians need to be aware of its presence and perform the transfer under ultrasound guidance to ensure the catheter bypasses the niche and enters the uterine cavity. Still the impact of c.s niche and its characteristics on outcome of ART is not clear.

ELIGIBILITY:
Inclusion Criteria:

* All women should have the following:

  * Aged from 18 - 37 years old.
  * Undergoing fresh ICSI cycles.
  * A normal uterus with no anomalies or pathologies.
  * At least one good-quality embryo/blastocyst available for transfer (3 BB and more according to Gardner and Schoolcraft grading system).
  * Easy mockup embryo transfer (i.e. the catheter is smoothly inserted without touching the fundus, no cervix tenaculum is used and the catheter is clean of blood).

Exclusion Criteria:

* Younger than 18 or older than 37 years old.
* Congenital uterine abnormality or pathology.
* Presence of a hydrosalpinx.
* Chronic diseases which are not suitable for pregnancy.
* ICSI cycles with fresh or frozen TESE samples.

Ages: 18 Years to 37 Years | Sex: Female
Age Groups: Adult
Study Population: It will be carried out in the department of Obstetrics and Gynecology, Zagazig University and in a private center.
Sampling Method: Non-Probability Sample
Enrollment: 266 (Estimated)
Dates: Start 2020-01-22 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
The Effect of cesarean section scar niche on ongoing pregnancy rate in ART cycles. | 2 years
  cesarean section scar niche will be measured by TVS

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig university, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Undecided